CLINICAL TRIAL: NCT01779284
Title: 24-Hour Efficacy of Travoprost/Timolol Benzalkonium Chloride BAK Free Compared With Latanoprost/Timolol Fixed Combination Therapy in Subjects With Open-Angle Glaucoma Insufficiently Controlled With Latanoprost Monotherapy
Brief Title: Travoprost/Timolol vs Latanoprost/Timolol Fixed Combination Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, AGP Konstas, Professor in Ophthalmology, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: A23
Record Dates: First submitted 2013-01-25; First posted 2013-01-30 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Glaucoma
Keywords: glaucoma; fixed combinations; 24-hour monitoring
MeSH Terms: conditions — Glaucoma | interventions — Travoprost; Latanoprost; Xalacom

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Travoprost/Timolol therapy (Active Comparator): Enrolled patients will be treated for 3 months with travoprost/timolol drops administered once in the evening. Evaluation of 24-hour pressure efficacy for this drug after 3 months of chronic therapy
  Interventions: Drug: Travoprost/timolol therapy; Drug: Latanoprost/Timolol therapy
- Latanoprost/Timolol therapy (Active Comparator): Enrolled patients will be treated for 3 months with travoprost/timolol drops administered once in the evening. 24-hour pressure monitoring will be carried out for this drug after 3 months of chronic dosing. All patients will be crossed over to therapy for 3 months with latanoprost/timolol fixed combination drops administered once in the evening. Evaluation of 24-hour pressure efficacy for this drug after 3 months of chronic therapy
  Interventions: Drug: Travoprost/timolol therapy; Drug: Latanoprost/Timolol therapy

INTERVENTIONS:
Drug: Travoprost/timolol therapy — Evaluation of 24-hour pressure efficacy with travoprost/timolol therapy after 3 months of chronic dosing
  Other Names: DuoTrav BAK Free
Drug: Latanoprost/Timolol therapy — Evaluation of 24-hour pressure efficacy for this drug after 3 months of chronic therapy
  Other Names: Xalacom

SUMMARY:
The primary objective of this crossover trial is to compare the 3-month, mean 24-hour intraocular pressure (IOP) control and safety obtained with two popular fixed combinations in glaucoma patients insufficiently controlled with latanoprost monotherapy. This study will compare the 24-hour efficacy of travoprost/timolol fixed combination without benzalkonium chloride given once in the evening, versus the latanoprost/timolol fixed combination given in the evening. It is assumed that travoprost/timolol fixed combination will provide better quality of 24-hour pressure control.

ELIGIBILITY:
Inclusion Criteria:

* Primary open-angle glaucoma or exfoliative glaucoma
* Patients who require additional IOP lowering on latanoprost monotherapy
* Morning IOP greater than 20 mm Hg on latanoprost monotherapy
* Untreated morning IOP greater than 26 mm Hg
* Patients older than 29 years
* Patients with early to moderate glaucoma (less than 14 decibel (dB) mean deviation visual field loss attributed to glaucoma and 0.8 or better vertical cup-to-disc ratio)
* On therapy with latanoprost monotherapy for at least 3 months
* Patients with a reliable visual field
* Best corrected distance Snellen visual acuity >1/10
* Corneal pachymetry within the 550 ± 50 μm range
* Patients should understand the study instructions
* Patients willing to attend all follow-up appointments and willing to comply with study medication usage
* Patients who have open, normal appearing angles

Exclusion Criteria:

* History of combined topical therapy
* Contraindication to prostaglandins or timolol
* History of ocular trauma or inflammation; intraocular surgery; severe dry eyes; use of contact lenses
* Sign of ocular infection except for mild blepharitis
* Any corneal abnormality that could have affected the measurement of IOP
* Chronic use of topical corticosteroids in the last 3 months before entering the study
* Current, or previous use of systemic corticosteroid treatment
* Uncontrolled systemic disease
* Change of a systemic medication during the study period
* Women of childbearing potential or lactating mothers
* Inability to understand the instructions and adhere to medications

Ages: 29 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Mean 24-hour intraocular pressure reduction between the two medications | 3 months
  Evaluation of 24-hour pressure every 4 hours at habitual position with calibrated Goldmann technology tonometer

SECONDARY OUTCOMES:
rate of adverse events with the two medications | 3 months
  At each visit local and systemic adverse effects that occurred during the treatment period will be recorded. Adverse events are evaluated by asking patients a general query about their state of health.
ocular surface indicators after 3 months of therapy with the two medications | 3 months
  Selected indicators (break up time of tears, Schirmer test and degree of corneal stain after application of fluorescein) will be employed after 3 months of therapy to determine the health status of ocular surface with the two medications.

CONTACTS AND LOCATIONS:
Locations (1):
- Glaucoma Unit, 1st University Department of Ophthalmology, Thessaloniki, Greece